CLINICAL TRIAL: NCT07390253
Title: Aflibercept 8mg in Patients Diagnosed With Neovascular Age-related Macular Degeneration (AMD) Who Have Been Treated With Aflibercept 2mg: the Eylea 8mg Switch Study. An Observational Study.
Brief Title: The Eylea 8mg Switch Study
Status: Active, not recruiting | Type: Observational
Sponsor: Vienna Institute for Research in Ocular Surgery (Other)
Responsible Party: Principal Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Principal Investigator, Vienna Institute for Research in Ocular Surgery
Other Study IDs: High Dose (HD) Eylea
Record Dates: First submitted 2026-01-28; First posted 2026-02-05 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Neovascular (Wet) Age-Related Macular Degeneration
Keywords: neovascular age-related macular degeneration; Aflibercept
MeSH Terms: conditions — Macular Degeneration | interventions — aflibercept

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- neovascular age-related macular degeneration (nAMD): Patient suffering from neovascular age-related macular degeneration (nAMD)
  Interventions: Drug: Aflibercept

INTERVENTIONS:
Drug: Aflibercept — Intravitreal injection with high dose (8 mg) aflibercept

SUMMARY:
This study will investigate if switching patients who appear to be sub-optimal responders to the current standard of care treatment with Aflibercept 2mg to Aflibercept 8mg will prolong treatment intervals and maintain visual acuity.

DETAILED DESCRIPTION:
Aflibercept 8 mg was recently approved by the European Medicines Agency (EMA) for the treatment of neovascular age-related macular degeneration (nAMD). The higher dosage promises prolongation of treatment intervals up to 16 weeks. Only limited clinical data is available on switching from so-called suboptimal or non-responders. A retrospective analysis showed that aflibercept in 3 mg or 4 mg doses can improve outcomes in patients who do not respond optimally to aflibercept 2 mg. It remains unclear whether switching to the above-mentioned and newly approved aflibercept 8 mg will prolong treatment intervals and stabilize visual acuity in patients who are not treatment-naive.

The present study is a single-center observational study. The plan is to include 50 eyes from 50 patients who have previously received aflibercept 2 mg injections. Patients receive a routine 8 mg aflibercept injection in the eye clinic based on the existing treat-extend regimen. At each visit, a visual acuity test, optical coherence tomography (OCT) imaging, and a standard slit lamp examination with fundoscopy are performed. The injection interval is extended by two weeks. If the two-week extension leads to deterioration, the interval is shortened by two weeks. Patients are monitored in the study for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients, who received prior intravitreal anti-VEGF-treatment for nAMD with Aflibercept 2mg. A minimum of four injections of Aflibercept 2mg is required. Therefore 16-24 weeks prior treatment with anti-VEGF is required in line with an interval of 4-8 weeks.
* Short treatment intervals of 4 or 8 weeks
* nAMD
* Age 21 or older
* Written informed consent

Exclusion Criteria:

* Chronic treatment with Bevacizumab or Faricimab
* Extensive macular fibrosis
* Diabetic retinopathy
* Other retinal pathologies (e.g. retinal vein occlusion)
* Dense media opacities (cataract, corneal scars)
* Vitreous hemorrhage
* Ocular or periocular infections
* Active intraocular inflammation
* Hypersensitivity to the active substance or to any of the excipients
* Prior Aflibercept 8mg treatment
* Pregnancy (for women in reproductive age a pregnancy test will be performed)

Ages: 21 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with neovascular AMD, which are suboptimal responders to the current standard of care
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-09-18 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Number of intravitreal injections | 12 months
  Total number of intravitreal injections will be assessed over 12 months

SECONDARY OUTCOMES:
corrected distance visual acuity (CDVA) | 12 months
  CDVA will be determined using ETDRS-charts in a distance of 4 metres and differences will be compared over a timeframe of up to 12 months
Central retinal thickness (CRT) | 12 months
  CRT will be assessed using optical coherence tomography (OCT) and will be compared up to 12 months
Intraretinal fluid (IRF) | 12 months
  IRF will be assessed using optical coherence tomography (OCT) and compared during a timeframe up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Findl, Prim. Prof. Dr., Principal Investigator — Vienna Institute for Research in Ocular Surgery
Locations (1):
- Vienna Institute for Research in Ocular Surgery, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided